CLINICAL TRIAL: NCT03411460
Title: Satisfaction of Using a Continuous Glucose Monitoring System to Monitor Interstitial Fluid Glucose Level in Hospitalized Insulin-dependent Diabetic Patients Treated Using a Portable Sub-cutaneous Pump
Brief Title: Satisfaction of Hospitalized Diabetic Patients Using a Continuous Glucose Monitoring System
Acronym: GLUCO FLASH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: logistical difficulties
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LOCAL/2016/MR-01
Record Dates: First submitted 2017-06-16; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2017-01

CONDITIONS: Insulin-Dependent Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interstitial glucose (Experimental): Glucose level tested by continuous monitoring device
  Interventions: Device: FreeStyle Libre™ system
- Blood glucose (Active Comparator): Glucose level tested on glucose monitor using standard finger prick
  Interventions: Procedure: Finger prick

INTERVENTIONS:
Device: FreeStyle Libre™ system — Measured non-invasively via scanner
  Arms: Interstitial glucose
Procedure: Finger prick — Blood test
  Arms: Blood glucose

SUMMARY:
The aim of the study is to establish whether routine usage of the FreeStyle Libre™ system (Abbott) improves satisfaction and quality of sleep in patients hospitalized for poor glycemic control with an indication for external insulin pump treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given their free and informed consent
* The patient must be insured or the beneficiary of an insurance policy
* The patient is aged at least 18 years and less than 75 years old.
* Patients have a BMI between 18 and 40kg/m2
* Diabetic patient admitted for glycemic instability with indication for treatment using an external insulin pump but otherwise in a stable clinical state

Exclusion Criteria:

* The subject is participating in another study
* The subject is in an exclusion period determined by a previous study
* The patients is under judicial protection or state guardianship
* The subject refuses to sign the consent form
* It proves impossible to give the subject clear information.
* The patient is pregnant, parturient or breastfeeding
* The patient is clinically unstable
* BMI less than 18 or over 40
* Existence of a severe rapidly progressive ischemic retinopathy or proliferative retinopathy.
* Serious psychiatric problems
* Chronic cutaneous infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
Satisfaction of patient-determined hospital care at discharge in the two groups | at discharge from hospital; maximum Day 5
  visual analogue scale 0-10

SECONDARY OUTCOMES:
Patient satisfaction concerning treatment for their diabetes | at discharge from hospital; maximum Day 5
  Diabetes Treatment Satisfaction Questionnaire
Patient quality of sleep | at each day of hospitalization and discharge; maximum Day 5
  Spiegel questionnaire
Satisfaction of nursing staff concerning care of patient | at end of study; maximum Day 5
  visual analogue scale response to 5 quesions
Time taken by nurse to measure circulating glucose level | Daily over length of hospitalization until maximum Day 5
  in minutes
Time necessary to achieve satisfactory equilibrium using insulin pump | maximum Day 5
  average daily glucose level < 1.50 g/l
Number of glucose readings above 2g/l and below 0.80g/l over the hospital stay | maximum Day 5
Number of hypoglycmic events with the corresponding glucose level | maximum Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No